CLINICAL TRIAL: NCT07396818
Title: A Trial of Kamlanoflast In Patients With Amyotrophic Lateral Sclerosis
Brief Title: Kamlanoflast In Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inflammasome Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFL-ALS-1004
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); ALS; Neuro-Degenerative Disease; Neuro-Degenerative Diseases; Motor Neuron Disease (MND)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Cohort A (Experimental): Low dose Kamlanoflast by oral administration
  Interventions: Drug: Kamlanoflast
- Dose Cohort B (Experimental): High dose Kamlanoflast by oral administration
  Interventions: Drug: Kamlanoflast

INTERVENTIONS:
Drug: Kamlanoflast — Low dose Kamlanoflast by oral administration
  Arms: Dose Cohort A
Drug: Kamlanoflast — High dose Kamlanoflast by oral administration
  Arms: Dose Cohort B

SUMMARY:
This is a study of Kamlanoflast in patients with ALS. Kamlanoflast is orally administered over 24 weeks. Its effects on inflammatory and functional parameters will be studied. Information on safety and tolerability will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of definite, probable, laboratory-supported probable, or possible ALS by revised El Escorial research criteria.
2. Ages 18 to 75 years.
3. Onset of weakness within three years of study enrollment.
4. ALS with progression, characterized either by:

i. a reduction of 0.5 points per month or greater on the ALS Functional Rating Scale-Revised (ALSFRS-R), which will be calculated based on (most recent ALSFRS-R at least 12 weeks from screening - ALSFRS-R at screening)/time interval; or ii. a calculated progression rate: (48 - ALSFRS-R at "time of diagnosis") / duration from onset to diagnosis (month) that is 0.5 points per month or greater.

e) Plasma NfL levels ≥ 2 times the upper limit of the age-specific reference values for normal at the measuring laboratory at screening.

f) Capable of providing informed consent. g) Capable and willing to follow study protocol. h) Ability to swallow pills and liquids at the time of the screening visit and, in the investigator's opinion have the ability to swallow for the duration of the study OR can be fed via a Gastrostomy (G) tube or Percutaneous Endoscopic capacity (PEG) tube.

i) Slow vital capacity (SVC) > 65% of predicted value for gender, height, and age (participants perform SVC for three trials and the best SVC will be used).

j) Females of childbearing potential must agree to abstain from sex or use adequate method of contraception for the duration of the study period and for 28 days after the last dose of study drug.

k) Males must agree to abstain from sex or use adequate method of contraception for the duration of the study period and for 28 days after the last dose of study drug.

l) If an approved therapy for ALS is used during the study, a steady dose must be used as follows: i. Participants who do not currently receive riluzole and do not plan to receive riluzole during the study period. Participants receiving riluzole are on a stable dose for at least 4 weeks before enrollment. Participants receiving riluzole are expected to remain on the same dose throughout the duration of the study.

ii. Participants who do not currently receive edaravone and do not plan to receive edaravone during the study period. Participants receiving edaravone must have completed at least 1 cycle of treatment before enrollment and are expected to continue edaravone treatment throughout the duration of the study.

Exclusion Criteria:

1. Inability to follow the study protocol, based on the investigator's assessment.
2. Pregnant or nursing women.
3. Recently（within 28 days）received other experimental treatments.
4. Presence of any active infections or inflammatory diseases at the time of enrollment that may confound the assessment of levels of inflammatory markers.
5. Taking any medication or supplements with anti-inflammatory effects, including but not limited to prednisone, colchicine, or curcumin.
6. Taking Qalsody (tofersen).
7. Taking any medications containing nucleotide reverse transcriptase inhibitors (NRTIs), including but not limited to Abacavir, Emtricitabine, Lamivudine, or Zidovudine; trade names Atripla, Biktarvy, Cimduo, Combivir, Complera, Delstrigo, Descovy, Dovato, Emtriva, Epivir, Epzicom, Genvoya, Odefsey, Retrovir, Stribild, Symfi, Symtuza, Triumeq, Trizivir, Truvada, Ziagen.
8. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant, according to investigator's judgment (e.g., cardiovascular instability, systemic infection), or clinically significant laboratory abnormality.
9. Clinically significant abnormal liver or kidney function at baseline (pre-dose). The following values [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN) or estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73m2] are exclusionary regardless of clinical symptoms.
10. Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent, in the investigator's opinion.
11. Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
12. Non-invasive ventilation, tracheostomy, oxygen supplementation for primary pulmonary pathology.
13. Current / anticipated need of diaphragm pacing system (DPS).
14. History of prior AAV gene therapy for any indication;
15. Presence of any clinically relevant diseases that, in the research team's opinion, would prevent the subject from completing the study, including but not limited to severe cognitive dysfunction or medical conditions other than ALS that affect physical function or life expectancy.
16. Plan to move away from the study site within the next 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | From drug initiation through study completion, an average of 28 weeks
  Safety: Defined as the occurrence of serious and non-serious treatment-emergent adverse events (TEAEs) and clinically significant treatment-emergent abnormalities in clinical and laboratory values, in ALS subjects treated with study treatment.
Incidence of Completing Study Treatment [Tolerability] | From drug initiation through study completion, an average of 24 weeks
  Tolerability: Defined as percentage of ALS subjects who complete the 24 weeks of study treatment (survival), without study drug-attributed intolerable AEs that lead to early permanent drug discontinuation.
Biological Efficacy | From enrollment through the end of study treatment at the Week 24 visit (longitudinal assessments)
  Biological Efficacy: Changes from baseline over 24 weeks (longitudinal assessments) in blood neuroinflammatory marker levels following oral study drug treatment.
ALS Functional Rating Scale Revised (ALSFRS-R) total and sub-domain scores | From enrollment to the end of study treatment at the Week 24 Visit (longitudinal assessments)
  Changes from baseline over 6 month period (longitudinal monthly assessments) in ALS Functional Rating Scale Revised (ALSFRS-R) total and sub-domain scores. The 12 domains included in the ALSFRS-R are rated on a 5-point scale, 0 to 4, with a maximum score of 48 indicating the highest level of functioning.
Slow vital capacity (SVC) | From enrollment to the end of study treatment at the Week 24 Visit (longitudinal assessments)
  Changes from baseline over 24 weeks in SVC (longitudinal assessments).

SECONDARY OUTCOMES:
Systemic Exposure | From enrollment to end of study treatment at the Week 24 Visit (longitudinal assessments)
  Systemic Exposure: Defined as blood study drug level measurement over 24 weeks of treatment (longitudinal assessments).

IPD SHARING:
Plan to Share IPD: No